CLINICAL TRIAL: NCT02760407
Title: A Randomized, Double-Blind, Parallel-Group, Placebo- and Active-Controlled, Multicenter Phase III Study of the Efficacy and Safety of Olokizumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Methotrexate Therapy
Brief Title: Evaluation of the Efficacy and Safety of Two Dosing Regimens of Olokizumab (OKZ), Compared to Placebo and Adalimumab, in Subjects With Rheumatoid Arthritis (RA) Who Are Taking Methotrexate But Have Active Disease
Acronym: CREDO 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Quintiles, Inc. (Industry); OCT Clinical Trials (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04041023
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate Rheumatoid Arthritis; severe Rheumatoid Arthritis; subcutaneous; Olokizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Olokizumab q4w (Experimental): Olokizumab 64 mg subcutaneous q4w +placebo+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular) in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
  Interventions: Drug: Olokizumab 64mg q4w; Drug: Placebo q2w
- Arm 2: Olokizumab q2w (Experimental): Olokizumab 64mg subcutaneous q2w + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Interventions: Drug: Olokizumab 64mg q2w
- Arm 3: Adalimumab q2w (Active Comparator): Adalimumab 40mg q2w subcutaneous + Methotrexate
  Subjects were administered adalimumab 40 mg q2w via SC injection as an active comparator+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Interventions: Drug: Adalimumab 40mg q2w
- Arm 4: Placebo q2w (Placebo Comparator): Placebo q2w subcutaneous + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
  Interventions: Drug: Placebo q2w

INTERVENTIONS:
Drug: Olokizumab 64mg q4w — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial
  Arms: Arm 1: Olokizumab q4w
Drug: Olokizumab 64mg q2w — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial
  Arms: Arm 2: Olokizumab q2w
Drug: Adalimumab 40mg q2w — 0.4 or 0.8 mL prefilled, single-dose syringe
  Other Names: Humira
  Arms: Arm 3: Adalimumab q2w
Drug: Placebo q2w — sodium chloride 0.9% solution supplied in either a 10 mL vial or ampoule, depending on market availability. Each placebo will be packed into a cardboard carton to contain 1 vial or ampoule
  Arms: Arm 1: Olokizumab q4w; Arm 4: Placebo q2w

SUMMARY:
The purpose of this study was to determine how effective and safe the study drug Olokizumab was in patients with Rheumatoid Arthritis (RA) who had been already receiving but not fully responding to treatment with methotrexate (MTX).

The primary objective of this study was to evaluate the efficacy of OKZ 64 mg administered subcutaneously (SC) once every 2 weeks (q2w) or once every 4 weeks (q4w) relative to placebo in subjects with moderately to severely active RA inadequately controlled by MTX therapy.

The secondary objective was to evaluate the efficacy of OKZ relative to adalimumab in subjects with moderately to severely active RA inadequately controlled by MTX therapy.

DETAILED DESCRIPTION:
The goal of this Phase III study was to assess the efficacy, safety and tolerability of OKZ in subjects with moderately to severely active RA who had responded inadequately to MTX. The primary endpoint of the trial was at Week 12. Olokizumab was expected to reduce the disease activity and improve physical function. The study was expected to provide safety information in a large group of subjects over at least a 24 week period.

This study included a 4-week Screening Period, a double-blind Treatment Period from Week 0 to Week 24, and a Safety Follow-Up Period from Week 24 to Week 44. Subjects were assessed for eligibility to enter the study during the 4-week Screening Period. A total of 1575 subjects were planned to be randomly assigned to 1 of 4 treatment groups in a 2:2:2:1 ratio (450, 450, 450, and 225 subjects per group, respectively):

1. Olokizumab 64 mg q4w: SC injection of OKZ 64 mg q4w (alternating with SC injection of placebo q4w to maintain blinding) + MTX
2. Olokizumab 64 mg q2w: SC injection of OKZ 64 mg q2w + MTX
3. Adalimumab 40 mg q2w: SC injection of adalimumab 40 mg q2w + MTX
4. Placebo: SC injection of placebo q2w + MTX

Throughout the double-blind Treatment Period, all subjects were required to remain on a stable dose of background MTX with a stable route of administration. Concomitant treatment with folic acid was required for all subjects. The last dose of study treatment (OKZ, adalimumab, or placebo) was at Week 22 in all groups.

Following Visit 2 (randomization; Week 0), subjects returned to the study site at least every 2 weeks through Week 24 for response and safety assessments.

At Week 14, subjects who had not improved by at least 20% in both swollen and tender joint counts were classified as nonresponders and were administered sulfasalazine and/or hydroxychloroquine as rescue medication in addition to the assigned treatment.

After completion of the 24-week double-blind Treatment Period, subjects either rolled over into the long-term open-label extension (OLE) study or entered the Safety Follow-Up Period. During the Safety Follow-Up Period, subjects returned for visits +4, +8, and +22 weeks after the last dose of study treatment.

Subjects who had discontinued randomized treatment prematurely were required to come for the End of Treatment (EoT) Visit 2 weeks after the last study treatment administration and then continue with the scheduled study visits.

Adverse events (AEs) were assessed throughout the study (starting when the subject signed the informed consent form) and evaluated using the Common Terminology Criteria for Adverse Events Version 4.0. There was ongoing monitoring of safety events, including laboratory findings, by the Sponsor or the Sponsor's designee. In addition, safety was assessed throughout the study by an independent Data Safety Monitoring Board and potential major adverse cardiac events were evaluated by an independent Cardiovascular Adjudication Committee.

The study was conducted at 208 sites across 18 countries globally (in US, European Union (EU),United Kingdom (UK), Russian Federation, Asia, Latin America).

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing and able to sign informed consent
* Subjects must have a diagnosis of adult onset RA classified by ACR/EULAR 2010 revised classification criteria for RA for at least 12 weeks prior to Screening. (If the subject was diagnosed according to ACR 1987 criteria previously, the Investigator may classify the subject per ACR 2010 retrospectively, using available source data)
* Inadequate response to treatment with oral, SC, or intramuscular MTX (defined as a subject with at least 12 weeks of exposure prior to Screening and with either absence of any documented clinically significant response, or documented initial clinical response with subsequent loss of that response or partial response) for at least 12 weeks prior to Screening at a dose of 15 to 25 mg/week (or ≥10 mg/week if intolerant to higher doses). The dose and route of administering MTX had to have been stable for at least 6 weeks prior to Screening. A lower dose of MTX (≥7.5 mg/week) was permitted for subjects enrolled in the Republic of Korea, consistent with local clinical practice.
* Subjects must be willing to take folic acid or equivalent throughout the study.
* Subjects must have moderately to severely active RA disease as defined by all of the following:

  * ≥6 tender joints (68 joint count) at Screening and baseline; and
  * ≥6 swollen joints (66 joint count) at Screening and baseline; and
  * CRP above the normal range (ULN) at Screening based on the central laboratory results.

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis or systemic rheumatic disease (eg, gout, psoriatic or reactive arthritis, Crohn's disease, Lyme disease, juvenile idiopathic arthritis, or systemic lupus erythematosus). However, subjects could have secondary Sjogren's syndrome or hypothyroidism.
* Subjects who are Steinbrocker class IV functional capacity (incapacitated, largely or wholly bed-ridden or confined to a wheelchair, with little or no self-care)
* Prior exposure to any licensed or investigational compound directly or indirectly targeting IL 6 or IL 6R (including tofacitinib or other Janus kinases and spleen tyrosine kinase [SYK] inhibitors)
* Prior treatment with cell depleting therapies including anti CD20 or investigational agents (e.g., CAMPATH, anti CD4, anti CD5, anti CD3, and anti CD19)
* Prior use of bDMARDs
* Use of parenteral and/or intra-articular glucocorticoids within 4 weeks prior to baseline
* Use of oral glucocorticoids greater than 10 mg/day prednisone (or equivalent) or change in dosage within 2 weeks prior to baseline
* Prior documented history of no response to hydroxychloroquine and sulfasalazine
* Prior use of cDMARDs (other than MTX) within the following windows prior to baseline (cDMARDs should not be discontinued to facilitate a subject's participation in the study, but should instead have been previously discontinued as part of a subject's medical management of RA):

  1. 4 weeks for sulfasalazine, azathioprine, cyclosporine, hydroxychloroquine, chloroquine, gold, penicillamine, minocycline, or doxycycline
  2. 12 weeks for leflunomide unless the subject has completed the following elimination procedure at least 4 weeks prior to baseline: Cholestyramine at a dosage of 8 grams 3 times daily for at least 24 hours, or activated charcoal at a dosage of 50 grams 4 times daily for at least 24 hours
  3. 24 weeks for cyclophosphamide
* Vaccination with live vaccines in the 6 weeks prior to baseline or planned vaccination with live vaccines during the study
* Participation in any other investigational drug study within 30 days or 5 times the terminal half-life of the investigational drug, whichever is longer, prior to baseline
* Other treatments for RA (e.g., Prosorba Device/Column) within 6 months prior to baseline
* Use of intra-articular hyaluronic acid injections within 4 weeks prior to baseline
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) on unstable dose or switching of NSAIDs within 2 weeks prior to baseline
* Previous participation in this study (randomized) or another study of OKZ
* Subjects with concurrent acute or chronic viral hepatitis B or C infection as detected by blood tests at Screening(e.g., positive for hepatitis B surface antigen [HBsAg], total hepatitis B core antibody [anti-HBc], or hepatitis C virus antibody [HCV Ab]). Subjects who are are positive for hepatitis B surface antibodies (anti-HBs), but negative for HBsAg and anti-HBc, will be eligible
* Subjects with human immunodeficiency virus (HIV) infection
* Subjects with:

  1. Suspected or confirmed current active TB disease or a history of active TB disease
  2. Close contact (i.e., sharing the same household or other enclosed environment, such as a social gathering place, workplace, or facility, for extended periods during the day) with an individual with active TB within 1.5 years prior to Screening
* Concurrent malignancy or a history of malignancy within the last 5 years (with the exception of successfully treated carcinoma of the cervix in situ and successfully treated basal cell carcinoma and squamous cell carcinoma not less than 1 year prior to Screening [and no more than 3 excised skin cancers within the last 5 years prior to Screening])
* Subjects with any infection requiring oral antibiotic or antiviral therapy in the 2 weeks prior to Screening or at baseline, injectable anti-infective therapy in the last 4 weeks prior to baseline, or serious or recurrent infection with history of hospitalization in the 6 months prior to baseline
* Subjects with evidence of disseminated herpes zoster infection, zoster encephalitis, meningitis, or other non-self-limited herpes zoster infections in the 6 months prior to baseline
* Subjects with planned surgery during the study or surgery ≤ 4 weeks prior to Screening and from which the subject has not fully recovered, as judged by the Investigator
* Subjects with diverticulitis or other symptomatic GI conditions that might predispose the subject to perforations, including subjects with history of such predisposing conditions (e.g., diverticulitis, GI perforation, or ulcerative colitis)
* Pre-existing central nervous system demyelinating disorders (e.g., multiple sclerosis and optic neuritis)
* History of chronic alcohol or drug abuse as judged by the Investigator
* Female subjects who are pregnant, currently lactating, have lactated within the last 12 weeks, or who are planning to become pregnant during the study or within 6 months of last dose of study treatment
* Female subjects of childbearing potential (unless permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 months of natural amenorrhea as defined by the amenorrhea with underlying status (e.g., correlative age) or 6 months of natural amenorrhea with documented serum follicle-stimulating hormone levels >40 mIU/mL and estradiol <20 pg/mL) who are not willing to use a highly effective method of contraception during the study and for at least 6 months after the last administration of study treatment OR Male subjects with partners of childbearing potential not willing to use a highly effective method of contraception during the study and for at least 3 months after the last administration of study treatment.
* Subjects with a known hypersensitivity to any component of the OKZ drug product, adalimumab, or placebo
* Subjects with a known hypersensitivity or contraindication to any component of the rescue medication
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1648 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (203):
- United States (64):
  - Arizona Arthritis & Rheumatology Associates, P.C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, El Cajon, California
  - MD Med Corp., Hemet, California
  - Valerius Medical Group, Los Alamitos, California
  - Rheumatology Center of San Diego, San Diego, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Pacific Arthritis Center Medical Grpoup, Santa Maria, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Center for Rheumatology Research, West Hills, California
  - Medvin Clinical Research, Whittier, California
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates LLC, Bridgeport, Connecticut
  - Javed Rheumatology Associates, Newark, Delaware
  - RASF - Clinical Research Center, Boca Raton, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Medical Research Center of Miami, Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - Arthritis Research, Palm Harbor, Florida
  - Family Clinical Trials, LLC., Pembroke Pines, Florida
  - AdventHealth Medical Group, PA, Tampa, Florida
  - Lovelace Scientific Resources, Inc., Venice, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Marietta Rheumatology Associates, PC, Marietta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Springfield Clinic, LLP, Springfield, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - The Arthritis & Diabetes Clinic, Inc., Monroe, Louisiana
  - Klein and Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - North MS Medical Clinics, Inc., Tupelo, Mississippi
  - Glacier View Research Instutute-Rheumatology, Kalispell, Montana
  - Physician Resrch Collaboration, Lincoln, Nebraska
  - Arthritis & Osteoporosis Associates, PA, Freehold, New Jersey
  - NYU Langone ambulatory care, Brooklyn, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - STAT Research, Inc., Dayton, Ohio
  - Clinical Research Source, Inc., Toledo, Ohio
  - Health Research of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Summerville, South Carolina
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, P.A., Austin, Texas
  - Accurate Clinical Management LLC, Baytown, Texas
  - Pioneer Research Solutions, Inc., Beaumont, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
  - Rheumatology Clinic of Houston, P.A., Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Accurate Clinical Mangemnt LLC, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Advanced Rheumatology of Houston, Houston, Texas
  - Accurate Clinical Research, Inc., League City, Texas
  - Endocrinology, Internal Medicine, Lubbock, Texas
  - Dr. Alex De Jesus Rheumatology, P.A., San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (15):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas-Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Medico CER, Quilmes, Buenos Aires
  - Clinica de Higado y Aparato Digestivo, Rosario, Santa Fe Province
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Institute Investigaciones Clinc Quilme, Buenos Aires
  - Atencion Integral en Reumatologia (AIR), Ciudad Autonoma Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - APRILLUS Asistencia e Investigacion, Ciudad Autonoma Buenos Aires
  - Instituto Centenario, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Instituto DAMIC Fundacion Rusculleda, Córdoba
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
- Brazil (14):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda., Curitiba, Paraná
  - Clinilive - Clínica do Idoso e Pesquisa Clínica, Maringá, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - LMK Serviços Médicos S/S Ltda, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, São Bernardo do Campo, São Paulo
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas Ltda., Rio de Janeiro
  - Clínica de Neoplasias Litoral, Santa Catarina
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo
  - Hospital Abreu Sodré - AACD, São Paulo
- Bulgaria (10):
  - UMHAT Pulmed OOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - Medizinski Zentar-1-Sevlievo EOOD, Sevlievo
  - MHAT - Shumen, AD, Shumen
  - NMTH "Tsar Boris III", Sofia
  - MHAT "Lyulin", EAD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - UMHAT Sv. Ivan Rilski EAD, Sofia
  - MC Synexus - Sofia EOOD, Sofia
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
- Colombia (5):
  - Centro de Investigacion Medico, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogotá
  - Medicity S.A.S., Bucaramanga
  - Clinica de Artritis Temprana S.A., Cali
- Czechia (18):
  - CCR Brno s.r.o, Brno
  - Revmatologie s.r.o., Brno
  - Nemocnice Jihlava p.o, Jihlava
  - MUDr. Gabriela Simkova ordinace lekare specialisty interna revmatologie, Kladno
  - CTCenter MaVe s.r.o., Olomouc
  - Vesalion s.r.o., Ostrava
  - Artroscan s.r.o., Ostrava - Trebovice
  - ARTHROHELP s.r.o., Pardubice
  - CCR Pardubice, Pardubice
  - Clintrial, s.r.o., Prague
  - Revmatologicky ustav, Prague
  - CCR Prague s.r.o., Prague
  - MUDR. Zuzana Urbanova Revmatologie, Prague
  - Affidea Praha, s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
  - MUDR. Zuzana URBANOVA Revmatologie, Praha 4 Nusle
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - PV Medical Services s.r.o., Zlín
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Medita Kliinik OÜ, Tartu
- Germany (6):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - Rheumapraxis Dr. med. Reiner Kurthen, Aachen, Westfalen
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
  - Studienambulanz Dr. Wassenberg, Northeim
- Hungary (8):
  - Principal SMO Kft., Baja
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Clinexpert Egeszsegugyi Szolg. es Ker. Kft., Budapest
  - Obudai Egeszsegugyi Centrum, Budapest
  - Kiskunhalasi Semmelweis Korhaz, Kiskunhalas
  - DRC Szekesfehervar, Székesfehérvár
  - MAV Korhaz és Rendelointezet, Szolnok
  - Vital Medical Center, Veszprém
- Dr.Saulite-Kandevica Private Practice, Liepāja, Latvia
- Lithuania (6):
  - Alytаus Regional S. Kudirkos Hospital, Public Institution, Alytus
  - Republican Kaunas Hospital, Public Institution, Kaunas
  - Klaipeda University Hospital, Public Institution, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Center Outpatient Clinic, Public Institution, Vilnius
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Mexico (11):
  - Centro de Investigacion Clínica GRAMEL S.C, México, DisMexicotrito Federal
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica SC, Guadalajara, Jalisco
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Clinicos Asociados BOCM S.C., Mexico City, Mexico City
  - Cryptex Investigacion Clinica S.C, Mexico City, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Clinical Research Institute S.C., México, State of Mexico
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City
- Poland (18):
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - MCBK Iwona Czajkowska Anna PodrażkaSzczepaniak S.C., Grodzisk Mazowiecki
  - Polimedica Centrum Badań, Profilaktyki I Leczenia, Kielce
  - Centrum Medyczne AMED, Lodz
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Szpital Wojewodzki im. Prymasa Kardynala Stefana Wyszynskiego, Sieradz
  - CCBR - Lodz - PL, Skierniewice
  - Clinmed Research, Skierniewice
  - RCMed, Sochaczew
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Samodzielny Publiczny ZOZ Tomaszow Lubelski, Tomaszów Lubelski
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Torun
  - Medycyna Kliniczna, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - McM Polimedica, Warsaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Zgierz
- Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Constanta, Constanța, Romania
- Russia (10):
  - Hospital n a Kuvatov, Ufa, Bashkortostan Republic
  - SPb SBHI "Clinical Rheumatological Hospital #25", Fourth Rheumatology Unit, Saint Petersburg, Leningradskaya Oblast'
  - FSBEI HE "FMSMU n.a. I.M. Sechenov of MoH of RF", University Hospital #2, Departament of New Drugs Introduction, Moscow, Moscovskaya Oblast
  - State Budgetary Healthcare Institution "City Clinical Hospital # 15 n.a O.M. Filatov" of Moscow Healtheare Department, Moscow, Moscow Oblast
  - SBHI of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a.Semashko", Nizhny Novgorod, Nizhny Novgorod Oblast
  - SBHI of Republic of Karelia "Republican Hospital named after V.A.Baranov", Petrozavodsk, Republic of Karelia
  - Non-govarnmental Healtheare Institution "Regional Clinical Hospital at Smolensk station of OJSC "Russian Railways", Smolensk, Smolensk Oblast
  - State Budgetary Healthcare Institution of Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg, Sverdlovsk Oblast
  - SBEI HPE "Ural State Medical University" of MoH of RF based MBI "Central City Clinical Hospital #6", Yekaterinburg, Sverdlovsk Oblast
  - Institute n a Nasonova, Moscow
- South Korea (6):
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - CHA Bundang Medical Center, Gyeonggi-do
  - Jeju National University Hospital, Jeju City
  - Severance Hospital, Yonsei University, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (2):
  - Chi Mei Medical Center, Tainan
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (6):
  - Torbay Hospital, Torquay, Devon
  - Whipps Cross University Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Maidstone Hospital, Maidstone, Kent
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, Merseyside

REFERENCES:
- [Derived] Smolen JS, Feist E, Fatenejad S, Grishin SA, Korneva EV, Nasonov EL, Samsonov MY, Fleischmann RM; CREDO2 Group. Olokizumab versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2022 Aug 25;387(8):715-726. doi: 10.1056/NEJMoa2201302. PMID 36001712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 208 clinical sites across 18 countries (US,EU,UK, Russian Federation, Asia, Latin America). 3359 subjects were screened and 1648 subjects were enrolled (randomized). A total of 1645 subjects were treated, and 1483 subjects completed the study. A total of 1648 subjects were analyzed for efficacy in the ITT Population and 1645 subjects were analyzed for safety in the Safety Population.
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64mg subcutaneous q4w + placebo + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.) + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
- Arm 2: Olokizumab q2w + Methotrexate: Olokizumab 64mg subcutaneous q2w + Methotrexate
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
- Arm 3: Adalimumab q2w + Methotrexate: Active Comparator, Adalimumab 40mg q2w subcutaneous + Methotrexate
  subjects were administered adalimumab 40 mg q2w via SC injection as an active comparator +concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 4: Placebo q2w + Methotrexate: Placebo subcutaneous q2w + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
Period: Overall Study
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Started | 479 | 464 | 462 | 243
Completed | 443 | 421 | 412 | 207
Not Completed | 36 | 43 | 50 | 36
Not completed — Death | 2 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 7 | 4 | 6
Not completed — Withdrawal by Subject | 25 | 31 | 37 | 25
Not completed — Violation of Eligibility criteria | 0 | 0 | 1 | 1
Not completed — Personal reasons | 0 | 0 | 0 | 1
Not completed — The subject was early discontinued due to lab Adverse Event as per Investigator's decision | 1 | 0 | 0 | 0
Not completed — Use of prohibited Medication | 0 | 0 | 1 | 0
Not completed — Subject didn't Completed Visits Schedule After Serious Adverse Event | 0 | 0 | 1 | 0
Not completed — Positive Quantiferon Testing, Patient Was Not Taken Prophylactic Medication | 1 | 0 | 0 | 0
Not completed — Investigator's Decision (Adverse Event) | 0 | 1 | 0 | 0
Not completed — Inadequately Enrolled | 0 | 0 | 0 | 1
Not completed — Withdrawal By PI's Decision | 0 | 1 | 0 | 0
Not completed — Subject Did not attend treatment period visits due to misunderstanding of protocol | 1 | 0 | 1 | 0
Not completed — Subject met permanent IP discontinuation criteria, did not agree for treatment period visits | 0 | 0 | 1 | 0
Not completed — Investigator recorded as Sponsor's decision - decreased lymphocyte level | 1 | 0 | 0 | 0
Not completed — Study Treatment Was Terminated At The Site | 0 | 0 | 1 | 0
Not completed — Subject Taken Out Of Study Due To Sponsor Investigating Investigational Product. | 1 | 0 | 0 | 0
Not completed — Inadequately enrolled patient refused to Follow-Up | 1 | 0 | 0 | 0
Not completed — Lack Of Efficacy Per PI | 0 | 0 | 0 | 1
Not completed — Patient had an upper respiratory infection and took medication that was not allowed | 1 | 0 | 0 | 0
Not completed — Investigator recorded as Adverse Event | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64mg subcutaneous q4w+ placebo+Methotrexate
  64 mg Olokizumab administered subcutaneously once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)+concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 3: Adalimumab q2w + Methotrexate: Active Comparator, Adalimumab 40mg q2w subcutaneous + Methotrexate
  Subjects were administered adalimumab 40 mg q2w via SC injection as an active comparator+ concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular)
- Total: Total of all reporting groups
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate | Total
Number analyzed (Participants) | 479 | 464 | 462 | 243 | 1648
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 389 | 379 | 367 | 192 | 1327
  >=65 years | 90 | 85 | 95 | 51 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.09) | 53.3 (11.92) | 54.3 (12.32) | 54.7 (11.85) | 53.9 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378 | 352 | 363 | 190 | 1283
  Male | 101 | 112 | 99 | 53 | 365
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 10 | 4 | 5 | 25
  Black or African American | 15 | 20 | 23 | 11 | 69
  White | 406 | 382 | 385 | 203 | 1376
  Other/Mixed | 52 | 52 | 50 | 24 | 178
Region of Enrollment [Number; unit: participants]
  Colombia | 18 | 17 | 16 | 8 | 59
  Argentina | 44 | 42 | 43 | 24 | 153
  Romania | 0 | 0 | 1 | 0 | 1
  Hungary | 15 | 13 | 13 | 10 | 51
  United States | 75 | 71 | 72 | 39 | 257
  Czechia | 58 | 50 | 51 | 30 | 189
  United Kingdom | 3 | 1 | 6 | 1 | 11
  Russia | 20 | 21 | 25 | 11 | 77
  Latvia | 1 | 3 | 0 | 0 | 4
  South Korea | 2 | 4 | 1 | 4 | 11
  Taiwan | 2 | 3 | 2 | 1 | 8
  Brazil | 33 | 33 | 30 | 16 | 112
  Poland | 90 | 85 | 87 | 46 | 308
  Mexico | 63 | 63 | 59 | 30 | 215
  Bulgaria | 18 | 20 | 19 | 8 | 65
  Lithuania | 22 | 22 | 22 | 8 | 74
  Germany | 11 | 13 | 10 | 6 | 40
  Estonia | 4 | 3 | 5 | 1 | 13
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.654 [16.96 to 52.74] | 28.656 [17.04 to 62.22] | 28.532 [17.48 to 56.52] | 28.573 [15.62 to 55.83] | 28.609 [15.62 to 62.22]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving American College of Rheumatology 20% (ACR20) Response
Description: The difference between OKZ and placebo in the percentage of subjects achieving an ACR20 response and remaining on randomized treatment and in the study at Week 12. (where a responder was defined as any subject satisfying ACR20 criteria and remaining on randomized treatment and in the study at Week 12) This endpoint served to demonstrate that the efficacy of OKZ was superior to placebo. American College of Rheumatology 20 % response is a composite defined as a ≥ 20% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥20% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: at Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64mg subcutaneous q4w+ placebo+Methotrexate
  64 mg Olokizumab administered subcutaneously once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w received placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.) + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 342 | 326 | 309 | 108
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The OKZ ACR20 response rate for the 64 mg q4w treatment group at Week 12 was expected to be at least 50% resulting in an expected difference in ACR20 response rates of 25 percentage points between the respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.270, 97.5% CI 2-sided [0.183 to 0.352]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The OKZ ACR20 response rate for the 64 mg q2w treatment group at Week 12 was expected to be at least 55%, resulting in an expected difference in ACR20 response rate of 30 percentage points between the respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.258, 97.5% CI 2-sided [0.171 to 0.341]

2. Secondary Outcome: Percentage of Subjects Achieving ACR20 Response: Olokizumab Comparison With Adalimumab
Description: A responder was defined as any subject satisfying ACR20 criteria and remaining on randomized treatment and in the study at Week 12.This endpoint served to demonstrate that the efficacy of OKZ was non-inferior to adalimumab, provided that superiority of adalimumab to placebo (assay sensitivity) was demonstrated concurrently based on the same endpoint.
  American College of Rheumatology 20 % response is a composite defined as a ≥ 20% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥20% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 342 | 326 | 309 | 108
Statistical Analysis 1: Comparison: Arm 3: Adalimumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The ACR20 response rate for adalimumab was expected to be at least 52.5% at Week 12; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.224, 95% CI 2-sided [0.148 to 0.298]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Adalimumab q2w + Methotrexate; A noninferiority margin of 12% was used for the comparison between OKZ and adalimumab with respect to this endpoint; Test type: Non-Inferiority — Non-Inferiority for each OKZ dosing regimen versus Adalimumab is achieved if the lower limit of the 97.5% confidence interval is greater than the protocol defined non-inferiority margin of -12%; Risk Difference (RD) = 0.045, 97.5% CI 2-sided [-0.022 to 0.112]
Statistical Analysis 3: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Adalimumab q2w + Methotrexate; A noninferiority margin of 12% was used for the comparison between OKZ and adalimumab with respect to this endpoint; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Risk Difference (RD) = 0.034, 97.5% CI 2-sided [-0.035 to 0.102]

3. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity
Description: Defined as Disease Activity Score 28-joint count (DAS28) C-reactive protein (CRP) <3.2, and remaining on randomized treatment and in the study at Week 12
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 220 | 210 | 177 | 31
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The DAS28 low disease activity (based on DAS28 [CRP] <3.2) response rate at Week 12 is estimated to be 10% in the placebo group and 22% in the 64 mg q4w OKZ group, resulting in an expected difference of 12 percentage points between respective OKZ group and placebo; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.332, 97.5% CI 2-sided [0.257 to 0.397]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The DAS28 low disease activity (based on DAS28 [CRP] <3.2) response rate at Week 12 is estimated to be 10% in the placebo group and 30% in the 64 mg q2w OKZ group, resulting in an expected difference of 20 percentage points between respective OKZ group and placebo; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.325, 97.5% CI 2-sided [0.250 to 0.391]

4. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity: Olokizumab Comparison With Adalimumab
Description: Percentage of subjects achieving low disease activity, defined as DAS28 (CRP) <3.2, and remaining on randomized treatment and in the study at Week 12; served to demonstrate that the efficacy of OKZ was noninferior to adalimumab, provided that superiority of adalimumab to placebo (assay sensitivity) was demonstrated concurrently based on the same endpoint
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 220 | 210 | 177 | 31
Statistical Analysis 1: Comparison: Arm 3: Adalimumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; The DAS28 low disease activity response rate for adalimumab was expected to be at least 27% at Week 12; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.256, 95% CI 2-sided [0.191 to 0.313]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Adalimumab q2w + Methotrexate; A noninferiority margin of 7.5% was used for the comparison between OKZ and adalimumab with respect to this endpoint; Test type: Non-Inferiority — Non-Inferiority for each OKZ dosing regimen versus Adalimumab is achieved if the lower limit of the 97.5% confidence interval is greater than the protocol defined noninferiority margin of -7.5%; Risk Difference (RD) = 0.076, 97.5% CI 2-sided [0.004 to 0.147]
Statistical Analysis 3: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Adalimumab q2w + Methotrexate; A noninferiority margin of 7.5% was used for the comparison between OKZ and adalimumab with respect to this endpoint; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; Risk Difference (RD) = 0.069, 97.5% CI 2-sided [-0.003 to 0.141]

5. Secondary Outcome: Improvement of Physical Ability From Baseline to Week 12, as Measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: Change of physical ability from baseline (the last available assessment prior to the first dose of the study treatment) to week 12, as measured by HAQ-DI. The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions.The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities, and each domain consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3 where 0 = without any difficulty (the best outcome), 1 = with some difficulty, 2 = much difficulty, and 3 = unable to do (the worst outcome). Each category is given a score by taking the maximum score of each question. A decrease from baseline indicates improvement for HAQ-DI.The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered. The HAQ-DI total score ranges from 0 (the best outcome) to 3 (the worst outcome).
Time Frame: Baseline to Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population. Subjects with a missing baseline are not included. Data after treatment discontinuation are Included, Data after discontinuing study are multiply Imputed based on the return to baseline assumption.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 473 | 449 | 456 | 235
score on a scale | -0.60 (0.028) | -0.65 (0.030) | -0.61 (0.029) | -0.42 (0.039)
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.19, 97.5% CI 2-sided [-0.29 to -0.09], Standard Error of Mean 0.046
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.22, 97.5% CI 2-sided [-0.33 to -0.12], Standard Error of Mean 0.046
Statistical Analysis 3: Comparison: Arm 3: Adalimumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Other; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.28 to -0.10], Standard Error of Mean 0.046

6. Secondary Outcome: Percentage of Subjects Achieving American College of Rheumatology 50% (ACR50) Response
Description: Difference between OKZ and placebo in the percentage of subjects achieving an ACR50 response and remaining on randomized treatment and in the study at Week 24
  American College of Rheumatology 50% Response is a composite defined as ≥50%, improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥50%, improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: at Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm 4: Placebo q2w + Methotrexate: Placebo subcutaneous q2w + Methotrexate
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral,subcutaneous,or intramuscular).
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 240 | 234 | 214 | 55
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.275, 97.5% CI 2-sided [0.192 to 0.349]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.278, 97.5% CI 2-sided [0.195 to 0.353]
Statistical Analysis 3: Comparison: Arm 3: Adalimumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Other; Risk Difference (RD) = 0.237, 95% CI 2-sided [0.165 to 0.303]

7. Secondary Outcome: Percentage of Subjects With Clinical Disease Activity Index (CDAI) ≤ 2.8 (Remission)
Description: Difference between OKZ and placebo in the percentage of subjects with Clinical Disease Activity Index (CDAI) ≤2.8 (remission) and remaining on randomized treatment and in the study at Week 24
Time Frame: at Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
Number analyzed (Participants) | 479 | 464 | 462 | 243
Participants | 58 | 51 | 60 | 10
Statistical Analysis 1: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p = 0.0003, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.080, 97.5% CI 2-sided [0.031 to 0.123]
Statistical Analysis 2: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Superiority; p = 0.001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.069, 97.5% CI 2-sided [0.020 to 0.111]
Statistical Analysis 3: Comparison: Arm 3: Adalimumab q2w + Methotrexate vs Arm 4: Placebo q2w + Methotrexate; Test type: Other; Risk Difference (RD) = 0.089, 95% CI 2-sided [0.046 to 0.127]

ADVERSE EVENTS:
Time Frame: All AEs were collected from the signature of the informed consent form until the last visit of the subject in the study (up to 22 weeks after the final dose of study treatment) regardless of relationship to study treatment, up to approximately 44 weeks. Any SAE with a start date after the Safety Follow-Up Period was not required to be reported unless the Investigator thought that the event might be related to either the study treatment, study treatment administration, or a protocol procedure
Description: All AEs and SAEs reported below are related to the Safety Population (safety population included all subjects who receive at least 1 dose of study treatment).
  Data for TEAEs were reported below. A Treatment Emergent Adverse Event (TEAE) is defined as an AE that started or worsened after the first dose of study treatment
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64mg subcutaneous q4w+ placebo+Methotrexate
  64 mg Olokizumab administered subcutaneously once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w will receive placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.) + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Adalimumab q2w + Methotrexate | Arm 4: Placebo q2w + Methotrexate
All-Cause Mortality (participants affected / at risk) | 2/477 | 3/463 | 1/462 | 1/243
Serious Adverse Events (participants affected / at risk) | 20/477 | 22/463 | 26/462 | 12/243
Other Adverse Events (participants affected / at risk) | 177/477 | 183/463 | 129/462 | 71/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Olokizumab q4w + Methotrexate (N=477) | Arm 2: Olokizumab q2w + Methotrexate (N=463) | Arm 3: Adalimumab q2w + Methotrexate (N=462) | Arm 4: Placebo q2w + Methotrexate (N=243)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 1 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratouveitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Olokizumab q4w + Methotrexate (N=477) | Arm 2: Olokizumab q2w + Methotrexate (N=463) | Arm 3: Adalimumab q2w + Methotrexate (N=462) | Arm 4: Placebo q2w + Methotrexate (N=243)
Nasopharyngitis (Infections and infestations) | 26 (34) | 29 (35) | 29 (32) | 18 (23)
Upper respiratory tract infection (Infections and infestations) | 29 (33) | 28 (31) | 26 (30) | 16 (17)
Urinary tract infection (Infections and infestations) | 14 (14) | 7 (9) | 19 (20) | 9 (10)
Bronchitis (Infections and infestations) | 10 (10) | 12 (12) | 11 (13) | 11 (11)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 20 (20) | 29 (29) | 6 (6) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 15 (15) | 25 (28) | 4 (4) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 (10) | 22 (24) | 5 (6) | 2 (2)
Alanine aminotransferase increased (Investigations) | 53 (88) | 41 (70) | 9 (20) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 24 (38) | 23 (27) | 8 (15) | 2 (2)
Hypertension (Vascular disorders) | 27 (31) | 25 (26) | 13 (13) | 8 (8)
Headache (Nervous system disorders) | 11 (12) | 10 (11) | 14 (17) | 12 (12)
Injection site erythema (General disorders) | 8 (8) | 8 (12) | 20 (51) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02760407/Prot_SAP_000.pdf